CLINICAL TRIAL: NCT05880459
Title: Comparison of Propofol-Nalbuphine and Propofol-Magnesium Sulphate Sedation for Patients Undergoing GIT Endoscopy
Brief Title: Sedation in Patients Undergoing GIT Endoscopy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noura Hasan Attia, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: ERCP
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Sedation for Patients Undergoing GIT Endoscopy
MeSH Terms: interventions — Propofol; Nalbuphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol and nalbuphine group (Active Comparator)
  Interventions: Drug: propofol and magnesium sulphate ,propofol and nalbuphine
- Propofol and magnesium sulfate group (Active Comparator)
  Interventions: Drug: propofol and magnesium sulphate ,propofol and nalbuphine

INTERVENTIONS:
Drug: propofol and magnesium sulphate ,propofol and nalbuphine — The patients will be randomly divided into 2 groups by using a computer-generated randomization tableAll patients will fast from solids for 8 h and from liquids for 2 h. After arrival at preoperative area an intravenous cannula will be placed in the peripheral vein of right hand for fluid infusion and medicine administration.
  All of the patients will be interviewed by the patient sedation satisfaction assessment tool (PSSI) regarding their experience 1 hour after the operation.

SUMMARY:
Comparison of propofol-nalbuphine and propofol-magnesium sulphate sedation for patients undergoing GIT endoscopy: a double-blind, randomized trial

DETAILED DESCRIPTION:
Endoscopy plays a significant role in the diagnosis and treatment of gastrointestinal diseases. Sedation has been used in clinical practice to make the procedure more comfortable, and improve patient satisfaction by helping patients rest during the procedure. (1) (2) The most common complications in gastrointestinal endoscopy are not related to the procedure, but are related to sedation; they include cardio-respiratory adverse events such as hypoxemia, hypoventilation, apnea, dysrhythmias, hypotension and vaso-vagal episodes (3).

Many studies have reported on use of propofol as a single agent for sedation during endoscopy. However propofol is often used in combination with another agent for other indications. The benefit of propofol in terms of shorter recovery and discharge times and higher patient satisfaction persists, when it is used in combination with other agents.

Propofol has limited analgesic effect and higher doses are often required, when it is used as a single agent for endonoscopy, resulting in higher sedation levels. Thus use of propofol in combination with other agents may be preferable to propofol alone. The combination may be easier to manage due to lower sedation levels and ability to reverse some of the sedation with the use of reversal agents for narcotics (4).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients scheduled for GIT endoscopy 2. Age 18-60 years old 3. ASA I-II. 4. BMI less than 30

Exclusion Criteria:

* 1. Heart disease (heart failure, angina, myocardial infarction, arrhythmia, etc.) 2. pulmonary disease (asthma, chronic obstructive pulmonary disease, pulmonary embolism, pulmonary edema, or lung cancer) 3. central nervous system abnormality 4. allergy to the study drugs 5. habitual sedative or analgesic use 6. pregnancy 7. Anticipated difficult airway.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The level of patient sedation | the time of endoscopy
  The level of patient sedation using Ramsay sedation agitation score (before induction of sedation (T0), 5 minutes after sedation (T1), 10 minutes after sedation (T2), and then every 30 minutes till complete recovery (T3, T4 and T5) to assess the depth of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abbas Youssef, Professor, Study Director — Assiut University; Ola Mahmoud Wahba, Assistant Professor, Study Director — Assiut University; Khaled Tolba Younes, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided
In the future

REFERENCES:
- [Background] Singh H, Poluha W, Cheung M, Choptain N, Baron KI, Taback SP. Propofol for sedation during colonoscopy. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD006268. doi: 10.1002/14651858.CD006268.pub2. PMID 18843709
- [Background] Rex DK, Khalfan HK. Sedation and the technical performance of colonoscopy. Gastrointest Endosc Clin N Am. 2005 Oct;15(4):661-72. doi: 10.1016/j.giec.2005.08.003. PMID 16278131
- [Background] Hinkelbein J, Lamperti M, Akeson J, Santos J, Costa J, De Robertis E, Longrois D, Novak-Jankovic V, Petrini F, Struys MMRF, Veyckemans F, Fuchs-Buder T, Fitzgerald R. European Society of Anaesthesiology and European Board of Anaesthesiology guidelines for procedural sedation and analgesia in adults. Eur J Anaesthesiol. 2018 Jan;35(1):6-24. doi: 10.1097/EJA.0000000000000683. PMID 28877145